CLINICAL TRIAL: NCT04045860
Title: The Effects of Complete Decongestive Therapy on Head and Neck Lymphedema in Post-surgical Head and Neck Cancer Patients (Randomized Control Trial)
Brief Title: Complete Decongestive Therapy on Head and Neck Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Our Lady of the Lake Hospital (Other)
Responsible Party: Principal Investigator, Leslie Son, Academic Research Director, Our Lady of the Lake Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDT for HNL
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Lymphedema of Face; Secondary Lymphedema
MeSH Terms: interventions — Observation

STUDY DESIGN:
Intervention Model Description: Randomized Control
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind randomization of patients and investigator outcome assessor. Patients that agree to participate will be randomized into a CDT treatment arm or a control arm that does not receive CDT. One speech pathologist on the study team will perform the CDT and will only be aware of the participant's cohort arm at the time of random assignment. The second speech pathologist will be blinded to the cohort arm and will be responsible for taking the cranio facial measurements for all participants to minimize investigator bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDT for head and neck lymphedema (Experimental): Complete Decongestive Therapy
  Interventions: Procedure: Complete Decongestive Therapy
- Standard of Care for head and neck lymphedema (Other): Observation
  Interventions: Other: Observation

INTERVENTIONS:
Procedure: Complete Decongestive Therapy — A combination of manual lymph drainage , compression bandaging, physical exercise and a skin care regimen
  Arms: CDT for head and neck lymphedema
Other: Observation — Standard of care is currently observation
  Arms: Standard of Care for head and neck lymphedema

SUMMARY:
This will be a prospective, randomized controlled study of ~60 adult patients who have undergone a laryngectomy, neck dissection, maxillectomy or mandibulectomy surgical procedure for the treatment of head and neck cancer at Our Lady of the Lake Hospital and have been referred by their physician for evaluation of head and neck lymphedema while serving as an inpatient. Consenting patients will be evaluated by certified speech and language pathologists trained to ascertain lymphedema severity using a series of visual and tangible measurements immediately following surgery and randomized into two cohorts, one receiving the complete decongestive therapy regimen and the other not receiving this specific combination treatment for their edema. Facial and neck measurements will be taken at baseline following surgery and at several points prior to and at discharge as well as at the 2 week follow up visit to the clinic. Measurements and overall change/reduction in edema will be compared between the cohorts.

DETAILED DESCRIPTION:
BACKGROUND:

Head and neck lymphedema (HNL) is a common and sometimes debilitating complication of head and neck cancer (HNC) treatment. It occurs when the lymphatic system is either overloaded or damaged and cannot clear the high protein lymphatic fluid within the interstitial tissues. This in turn causes inflammation, connective tissue proliferation and overall functional impairment of the lymph system and bodily extremities. The long-term effects that edema can have in the cranio-facial region are not simply a cosmetic nuisance, but can lead to severe functional and psycho-social issues when affecting the lips, tongue, throat, eyes, mouth and neck. The ability to communicate, swallow, breath and see can be greatly impeded by the lymphatic swelling, which clearly affects the quality of life for many patients. Additional deficits may include dysfunction of the arms and shoulders with reduced cervical range of motion. Although lymphedema is well recognized in patients within the fields of urinary, breast and gynecologic cancer, it has only recently been addressed in the area of head and neck cancer.

The therapeutic management of HNL in HNC patients is a growing topic of research, as this condition pushes to the forefront and crosses over multi-disciplinary departments from otolaryngology to cancer therapy to speech and language therapy and rehabilitation. Historically, the technique of manual lymph drainage (MLD), a series of gentle circular massage strokes applied to the skin to increase lymphatic flow has been used. Decades later, the MLD technique was combined with compression bandaging, physical exercises and a skin care regiment to create a complete decongestive therapy (CDT) in the outpatient setting and is now considered to be best practice for outpatient lymphedema treatment at some institutions. The HNL program at M.D. Anderson Cancer Center has also created a series of formal evaluation and treatment techniques which include patient interviews/survey, visual assessment of the cranio-facial, neck and shoulder areas, functional assessments of communication and swallowing, photography, tape measurements and staging scales of edema to characterize the appearance and severity of the swelling.

Herein, investigators propose to examine the effects of complete decongestive therapy on head and neck cancer patients at Our Lady of the Lake Regional Medical Center who experience post-surgical head and neck lymphedema after total laryngectomy, neck dissection, maxillectomy or mandibulectomy compared to a control cohort. Investigators aim to assess the improvement of patient outcomes through the use of this technique to reduce cranio-facial edema and compare to those who do not receive CDT in an in-patient setting. Our study is novel in that there is minimal data on the effect of CDT in the acute care setting and in the areas of the head and neck, hence contributing to the growing body of knowledge about this therapy in this acute patient population.

OBJECTIVES:

The objective of of this research study is to assess physical improvements in visual, measureable and functional outcomes in head and neck cancer patients with head and neck lymphedema who have undergone Complete Decongestive Therapy (CDT) as a part of in-patient care at Our Lady of the Lake Hospital and compare this to patients in a control group who do not receive CDT.

STUDY DESIGN:

This will be a prospective, randomized controlled study of ~60 adult patients who have undergone a laryngectomy, neck dissection, maxillectomy or mandibulectomy surgical procedure for the treatment of head and neck cancer and have been referred by their physician for evaluation of head and neck lymphedema while admitted to inpatient care at Our Lady of the Lake Regional Medical Center following surgery. Patients will be evaluated by certified speech and language pathologists trained to ascertain lymphedema severity using a series of visual and tangible measurements immediately following surgery. Specific therapies for speech and language performance are provided beginning 24-72 hours post op per standard of care. At the time of speech therapy, patients will be informed and consented at the hospital bedside about this study. Those that agree to participate will be randomized into a CDT treatment arm or a control arm. The CDT therapy arm will be a combination of manual lymph drainage (MLD), tissue compression or kinesio tape bandaging, remedial exercises and a skin care regiment. This therapy will be administered every time the patient is seen by the speech pathologist, which is typically on a daily basis until discharge. Patients who are randomized into the control arm will not receive the specific CDT, but will still receive any speech or language therapy or other medical treatment services that are standard for their care management plan. Cranio-facial measurements will be taken of both cohorts by a blinded measurer prior to therapy and prior to hospital discharge, after several rounds of CDT have been administered to the patient. Those in the non-CDT cohort will be measured at the day of inpatient consult and again on day of discharge. Changes in the measurements will determine if the CDT has a positive effect on the edema symptoms.

One speech pathologist on the study team will perform the CDT or control therapy and will only be aware of the participant's cohort arm at the time of random assignment. A second speech pathologist will be blinded to the cohort arm and will be responsible for taking the cranio facial measurements for all participants.

Patients will be randomized into one of two groups. Group A will receive the CDT during their inpatient stay. Group B will not receive the CDT. The randomization of the patients into these 2 cohorts will be predetermined by pulling 15 permuted blocks of 4 (Ex. AABB, ABAB, BABB, ABBA, etc) pre-drawn by an individual not involved in the therapy. The permuted blocks will be lined up sequentially (Ex. AABBABABBABBABBA…..) and each letter placed in one of 60 envelopes. The speech pathologist assigned to the patient will pull the next envelope in order to determine if the patient will be in Group A (CDT) or Group B (no CDT) post-surgery. The principal investigator and the individual who will perform the measurements will be completely blinded to the patient's cohort assignment and in this way, minimize investigator bias.

A medical chart review will also be conducted to gather additional variables such as age, gender, race and any prior head and neck cancer medical history.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older)
* Any head and neck cancer patient undergoing laryngectomy, neck dissection, maxillectomy or mandibulectomy
* Inpatient and referred for HNL treatment following surgery
* Patients with previous chemoradiation therapy or head and neck surgery accepted

Exclusion Criteria:

* Patients under the age of 18 years of age
* Patients who undergo neck dissection surgery that do not present with symptoms of HNL
* Patients with free tissue transfer reconstruction
* Unwilling or unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in composite facial measurements | During inpatient stay, approximately 3-4 days
  2 % percent change of composite facial measurement

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Mays, MD, Principal Investigator — Our Lady of the Lake
Locations (1):
- Our Lady of the Lake Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified upon collection